CLINICAL TRIAL: NCT01196689
Title: An Open, Single Centre, Phase I Study in Male Adolescents With Asthma, Aged 12 to 17 Years, to Assess Pharmacokinetics of Orally Administered AZD1981 Tablets 100 mg Twice Daily for 61/2 Days
Brief Title: Pharmacokinetics in Adolescents
Acronym: PEAK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Medical Science Director (MSD), AstraZeneca
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D9830C00021
Record Dates: First submitted 2010-08-31; First posted 2010-09-08 (Estimated); Last update posted 2011-03-07 (Estimated); Status verified 2011-03

CONDITIONS: Asthma
Keywords: Pharmacokinetics AZD1981; Asthma
MeSH Terms: conditions — Asthma | interventions — AZD1981

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): AZD1981 100 mg twice daily for 6 ½ days
  Interventions: Drug: AZD1981 100 mg twice daily for 61/2 days

INTERVENTIONS:
Drug: AZD1981 100 mg twice daily for 61/2 days — 100 mg tablets

SUMMARY:
The purpose of this study is to study pharmacokinetics in adolescents.

DETAILED DESCRIPTION:
An open, single centre, phase I study in male adolescents with asthma, aged 12 to 17 years, to assess pharmacokinetics of orally administered AZD1981 tablets 100 mg twice daily for 61/2 days.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* A minimum of 6 months documented history of asthma
* Be a non-smoker or ex-smoker who has stopped smoking for >6 months prior to Visit 1 (pre-entry)

Exclusion Criteria:

* Any clinically significant disease or disorder which, in the opinion of the investigator, may either put the patient at risk because of participation in the study, or influence the result of the study, or the patient's ability to participate
* Any clinically relevant abnormal findings in phys.examination, clinical chemistry, haematology, urinalysis, vital signs, or ECG at baseline which, in the opinion of the investigator, may put the patient at risk because of his participation in the study

Ages: 12 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2010-10; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
The primary steady-state outcome variables to assess systemic exposure and oral clearance will be AUCτ, Css,max, Css,trough, and CL/F of AZD1981 | 0 hours after last dose
The primary steady-state outcome variables to assess systemic exposure and oral clearance will be AUCτ, Css,max, Css,trough, and CL/F of AZD1981 | 0.5, hours after last dose
The primary steady-state outcome variables to assess systemic exposure and oral clearance will be AUCτ, Css,max, Css,trough, and CL/F of AZD1981 | 1 hour after last dose
The primary steady-state outcome variables to assess systemic exposure and oral clearance will be AUCτ, Css,max, Css,trough, and CL/F of AZD1981 | 3 hours after last dose
The primary steady-state outcome variables to assess systemic exposure and oral clearance will be AUCτ, Css,max, Css,trough, and CL/F of AZD1981 | 4 hours after last dose
The primary steady-state outcome variables to assess systemic exposure and oral clearance will be AUCτ, Css,max, Css,trough, and CL/F of AZD1981 | 6 hours after last dose
The primary steady-state outcome variables to assess systemic exposure and oral clearance will be AUCτ, Css,max, Css,trough, and CL/F of AZD1981 | 8 hours after last dose
The primary steady-state outcome variables to assess systemic exposure and oral clearance will be AUCτ, Css,max, Css,trough, and CL/F of AZD1981 | 12 hours after last dose

SECONDARY OUTCOMES:
Tolerability and safety assessed by adverse events | During 7 days
Efficacy assessed by Forced Expiratory Volume (FEV) in one second and Asthma Control Questionnaire | Day 1 and 7

CONTACTS AND LOCATIONS:
Overall Officials: Christer Hultquist, Study Director — AstraZeneca
Locations (1):
- Research Site, Uppsala, Uppsala County, Sweden